CLINICAL TRIAL: NCT07044739
Title: The Effect of Information on the Use of Anti-embolic Stockings on Discharge Readiness and Satisfaction With Nursing Care in Patients Undergoing Vein Surgery
Brief Title: Information on the Use of Anti-embolic Stockings in Patients Undergoing Vein Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Ezgi Arslan, PhD, Research Assisstant (Principal Investigator), Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Use of Anti-embolic Socks
Record Dates: First submitted 2025-06-13; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-05

CONDITIONS: Nursing Care; Vascular Surgery; Patient Education
Keywords: nursing care; vascular surgery; discharge; postoperative period

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training on the use of anti-embolic stockings (Experimental): Information will be provided on the use of anti-embolic stockings. During the information session, an educational material titled "Use of Anti-Embolic Stockings" will be prepared by the researcher for the patients. The content of the training will be created to cover the purpose of using anti-embolic stockings, how to use them, and the points to be considered during use. The training is expected to take approximately 20 minutes. The training will be given face-to-face in the patient room by the researcher. The created training material will be evaluated in terms of content and form by 1 specialist in the field of Cardiovascular Surgery and 4 specialists in the field of Surgical Diseases Nursing using the "Nursing Education Material Evaluation Tool" (HEMDA) and expert opinions will be obtained. The content of the training material will be finalized in line with the opinions received.
  Interventions: Behavioral: Patient Education on the Use of Anti-Embolic Stockings
- Usual care (No Intervention): Control group patients will receive routine nursing care in the clinic.

INTERVENTIONS:
Behavioral: Patient Education on the Use of Anti-Embolic Stockings — The researcher will provide verbal information to the patients with the educational material titled "Use of Anti-Embolic Stockings", the stages of wearing anti-embolic stockings will be shown to the patients, and the educational material will be left next to the patients in the intervention group. The educational content covers the purpose of using anti-embolic stockings, how to use them, and the points to be considered during use.
  Arms: Training on the use of anti-embolic stockings

SUMMARY:
The aim of this study was to investigate the effect of information given to patients undergoing vein surgery regarding the use of anti-embolic stockings on their readiness for discharge and satisfaction with nursing care.

DETAILED DESCRIPTION:
Today, with the widespread use of evidence-based practices in nursing care, it is recommended that mechanical prophylaxis methods be widespread in preventing venous thromboembolism in patients. In particular, evaluating whether the clinical presentations of patients are suitable for these methods, applying mechanical prophylaxis safely and effectively, and informing patients about the subject for the home care process are among the basic responsibilities of nurses. The nurse who will provide the training should know all the practices that the patient will perform on how to care for himself/herself at home, explain them to the patient in an appropriate language, and first demonstrate them in person. Before providing training, nurses should provide training after passing a scale. The cheapest, most accessible and most frequently applied method among mechanical prophylaxis methods is the use of anti-embolic stockings, also known as elastic stockings. Elastic pressure stockings are widely used in the postoperative period. These stockings are effective by reducing endothelial damage, venous stasis and hypercoagulation processes that are effective in the emergence of venous thromboembolism. Before using these stockings, it is also the responsibility of the nurses to evaluate whether the patients have a possible allergy related to the stockings or a disease such as neuropathy or arterial insufficiency that would prevent the use of the stockings, to inform the patient about important points such as using the stockings individually, to be suitable for the person's leg size, to be wrinkle-free when worn or to be worn while lying down with the feet elevated, and to monitor the negative effects such as ischemia, numbness, and injuries that may occur during the use process. The nurse should be proactive in informing the patient about the use of anti-embolic stockings, which is one of the mechanical methods used to prevent venous stasis after vein surgery in patients, to ensure that they use them correctly, and to motivate the patient. In this context, the patient should be well informed in order to support the use of anti-embolic stockings at home starting from the post-operative period and to maintain compliance. The information headings should cover the purpose of anti-embolic stockings, frequency of use, and things to consider during use. No study has been found in the literature regarding the use of anti-embolic stockings in patients undergoing vein surgery, and it is thought that this study will increase the readiness for discharge and satisfaction levels of patients undergoing vein surgery by informing them.

ELIGIBILITY:
Inclusion Criteria:

• Having had vein surgery

Exclusion Criteria:

* Having hearing/vision/mental problems
* Having been diagnosed with a psychological illness (schizophrenia, depression)
* Having any of the contraindications for the use of anti-embolic stockings in the patient (the patient has peripheral arterial disease or bypass grafts, peripheral neuropathy or other causes of sensory impairment, heart failure, pulmonary or leg edema, poor skin condition due to dermatitis/diabetes/venous ulcers, allergy or sensitivity to the materials in the stockings, and leg deformities that prevent the stockings from fitting properly)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Readiness for Discharge | Immediately after the intervention
  Readiness for discharge will be assessed with the Discharge Readiness Scale. : The scale consists of 8 questions and 4 sub-dimensions as personal status, knowledge, coping, and expected support. The questions in the scale are assessed between '0=not ready' and '10=completely ready'. A total of 0-80 points can be obtained from the scale according to the answers given to the questions, and an increase in the score indicates that the level of readiness of the patients for discharge increases. In the scale dimension scores, a score of 7 and above is assessed as the patient is ready for discharge, and a score below 7 is assessed as not ready for discharge.
Nursing care satisfaction | Immediately after the intervention
  Nursing care satisfaction will be assessed with the Nursing Care Satisfaction Scale. The 19 items in the scale are 5-point Likert type and aim to define patients' satisfaction with various aspects of nursing care. The scoring used to determine the degree of satisfaction includes the following statements: 1- Not at all satisfied, 2- Rarely satisfied, 3- Satisfied, 4- Very satisfied, 5- Completely satisfied. The scale has no cut-off point. The patient's satisfaction with nursing care is assessed with the scale as long as the patient stays in the patient's room. The score evaluation is made on a 0-100 score by adding the scores of all items on the scale and converting them to 100. It is reported that a total score of 100 indicates satisfaction with all aspects of nursing care. A high total score also indicates high patient satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Ezgi Arslan, PhD, Principal Investigator — Aydin Adnan Menderes University

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author or reasonable request.
Supporting Information: CSR
Time Frame: 12 months after publication
Access Criteria: Relevance to the topic of the study and approval of all-authors within 1 month of receiving the request.